CLINICAL TRIAL: NCT03007979
Title: A Phase II Clinical Trial Assessing the Safety of an Alternative Dosing Schedule of Palbociclib in Metastatic Hormone Receptor Positive Breast Cancer
Brief Title: Alternative Dosing Schedule of Palbociclib in Metastatic Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201612098
Record Dates: First submitted 2016-12-19; First posted 2017-01-02 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Breast Carcinoma; Cancer of Breast; Malignant Tumor of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole; Fulvestrant; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib + letrozole or + fulvestrant (Experimental): * Palbociclib should be taken by mouth with food on a 5 days on/2 days off schedule (meaning: on Days 1-5, 8-12, 15-19, and 22-26 of each 28-day cycle).
  * Patients who are receiving letrozole will take it daily by mouth, every day of each 28-day cycle.
  * Patients who are receiving fulvestrant will receive it as two intramuscular injections (one into each buttock) on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter.
  * Goserelin is given as a subcutaneous injection every 28 days. It is preferred to be given on Day 1 of each cycle, but it may be administered on any day of the treatment cycle to accommodate its specific Q28-day cycle. It will be given to pre- or peri-menopausal women only.
  * Optional research biopsy at baseline and progression
  * Blood for research at baseline, cycle 1 day 15, cycle 2 day 1, every 2-3 months (to coincide with imaging studies), and time of progression
  Interventions: Drug: Palbociclib; Drug: Letrozole; Drug: Fulvestrant; Procedure: Optional research biopsy; Drug: Goserelin; Procedure: Research blood draw; Procedure: Circulating tumor cell blood draw; Procedure: Tumor biopsy (optional)

INTERVENTIONS:
Drug: Palbociclib — Palbociclib at a dose of 125 mg should be taken by mouth with food on a 5 days on/2 days off schedule
  Other Names: Ibrance
Drug: Letrozole — Patients who are receiving letrozole will take it daily by mouth, every day of each 28-day cycle, at a dose of 2.5 mg.
  Other Names: Femara
Drug: Fulvestrant — Patients who are receiving fulvestrant will receive it at a dose of 500 mg as two 5 mL intramuscular injections (one into each buttock) on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter.
  Other Names: Faslodex
Procedure: Optional research biopsy — Patients may consent to paired tumor biopsies at baseline and time of progression.
Drug: Goserelin — Goserelin is given as a subcutaneous injection every 28 days. It is preferred to be given on Day 1 of each cycle, but it may be administered on any day of the treatment cycle to accommodate its specific Q28-day cycle. It will be given to pre- and peri-menopausal women only.
  Other Names: Zoladex
Procedure: Research blood draw — -Blood will be drawn at the following time points for serum, plasma, cfDNA, and germline DNA (only at baseline):
  * Baseline
  * C1D15
  * C2D1
  * Every 2-3 months thereafter (to coincide with imaging studies)
  * Time of progression
Procedure: Circulating tumor cell blood draw — -Baseline, cycle 2 day 1, post 2 or 3 months of therapy (to coincide with first tumor imaging), and progression
Procedure: Tumor biopsy (optional) — -Baseline and progression

SUMMARY:
The investigators propose to conduct a study to test an alternative dosing schedule of palbociclib. With the current three-week on and one week off schedule, a significant number of patients develop grade 3 or higher degree of neutropenia and require dose reduction and sometimes discontinuation. This potentially compromises the efficacy of the drug. In addition, as the half-life of palbociclib is 27 hours, 1 week break with the standard 3 weeks on and 1 week off dosing schedule could potentially lead to recovery of Rb phosphorylation during the off week. Hence, the investigators propose a 5 days on and 2 days off schedule each week without any weeks off drug. Although the cumulative doses each 28-day cycle is roughly the same with this schedule compared to conventional dosing, the bone marrow is not exposed to the drug continuously for 21 days and rather gets frequent breaks from therapy. The investigators hypothesize that the 5 days on and 2 days off schedule is more tolerable with less frequent high grade neutropenia and dose interruption/reduction. In addition, this schedule also provides for a more continuous drug delivery to the patient since there is not a week's break in therapy, which could ultimately prove to be more efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic ER+ and/or PR+ and HER2- breast cancer who are candidates for palbociclib in combination with either letrozole or fulvestrant per treating physician.
* Presence of measurable or non-measurable disease by RECIST 1.1 criteria.
* One prior systemic therapy in the metastatic setting is allowed, but patients who have not had any prior systemic therapies in the metastatic setting are also eligible.

  *Note: patients who were started on endocrine therapy monotherapy as their 1st line or 2nd line systemic therapy in the metastatic setting for no more than 28 days and without clinical progression prior to the initiation of the study drug therapy are allowed to enroll on the study as their 1st line or 2nd line therapy, respectively.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
* Total bilirubin ≤ institutional upper limit of normal (IULN) or total bilirubin ≤ 3.0 x IULN with direct bilirubin within normal range in patients with documented Gilbert's syndrome
* AST(SGOT)/ALT(SGPT) ≤ 1.5 x IULN (up to 5 x IULN in patients with liver disease)
* Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with serum creatinine levels above institutional normal (calculated by Creatinine Clearance Estimate by Cockcroft-Gault Equation)
* Pre- or post-menopausal women are allowed. If pre- or peri-menopausal, concurrent ovarian suppression for pre- or peri-menopausal women is required.
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to swallow and retain oral medication.
* Washout of at least 3 weeks from prior chemotherapy or targeted therapy that induces myelosuppression and recovery of treatment related adverse events to grade 1 or less, with the exception of alopecia, is required prior to the start of palbociclib.
* Ability to understand and willingness to sign an Institutional Review Board (IRB) approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior therapy with any CDK inhibitor.
* Currently receiving any other investigational agents.
* Currently receiving exogenous estrogen replacement (topical vaginal estrogen therapy is allowed).
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis which could affect the evaluation of all-cycle adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib or other agents used in the study.
* Receiving any medications or substances that are potent inhibitors or inducers of CYP3A isoenzymes within 7 days prior to registration.
* Clinically significant history of liver disease.
* A condition that would interfere with enteric absorption.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with palbociclib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia X Ma, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krishnamurthy J, Luo J, Suresh R, Ademuyiwa F, Rigden C, Rearden T, Clifton K, Weilbaecher K, Frith A, Roshal A, Tandra PK, Cherian M, Summa T, Haas B, Thomas S, Hernandez-Aya L, Bergqvist M, Peterson L, Ma CX. A phase II trial of an alternative schedule of palbociclib and embedded serum TK1 analysis. NPJ Breast Cancer. 2022 Mar 21;8(1):35. doi: 10.1038/s41523-022-00399-w. PMID 35314693
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Started | 55
Completed | 54
Not Completed | 1
Not completed — Deemed not eligible prior to starting palbociclib | 1

BASELINE CHARACTERISTICS:
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 61 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Rate of Grade 3 or Higher Neutropenia
Description: * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
  * Grade 3 neutropenia: <1000-500/mm^3; <1.0-0.5 x 10e9/L
  * Grade 4 neutropenia: <500/mm^3; <0.5 x 10e9/L
Time Frame: Through the first 29 days of treatment
Population: The following participants were not evaluable for this outcome measure: 4 participants did not take palbociclib dose as per protocol and were without dose-limiting toxicity; 2 participants withdrew in cycle 1, and 1 participant went off treatment in cycle 1 due to adverse events unrelated to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 47
Participants | 10

2. Secondary Outcome: Rate of Grade 3 or Higher Neutropenia
Description: as for outcome 1
Time Frame: Through 30 day follow-up (estimated to be 25 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 47
Participants | 23

3. Secondary Outcome: Rate of Palbociclib Dose Reduction
Description: -Percentage of participants who have a palbociclib dose reduction during treatment
Time Frame: Through the completion of treatment (estimated to be 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
Participants | 13

4. Secondary Outcome: Rate of Palbociclib Dose Interruption
Description: -Percentage of participants who have a palbociclib dose interruption during treatment
Time Frame: Through the completion of treatment (estimated to be 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
Participants | 39

5. Secondary Outcome: Rate of Palbociclib Discontinuation
Description: -Percentage of participants who discontinue palbociclib due to adverse event
Time Frame: Through the completion of treatment (estimated to be 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
Participants | 2

6. Secondary Outcome: Adverse Event Profile of Palbociclib
Description: * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
  * Relationship of possible, probably, or definitely related.
Time Frame: Through the 30 day follow-up (estimated to be 25 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
Participants
  Grade 1-2 anemia | 31
  Grade 3-4 anemia | 4
  Grade 1-2 blurred vision | 1
  Grade 1/2 constipation | 5
  Grade 1-2 diarrhea | 8
  Grade 1-2 dyspepsia | 1
  Grade 1-2 gastric ulcer | 1
  Grade 1-2 mucositis oral | 11
  Grade 1-2 nausea | 16
  Grade 1-2 oral dysesthesia | 1
  Grade 1-2 vomiting | 7
  Grade 1-2 chills | 3
  Grade 1-2 fatigue | 22
  Grade 1-2 fever | 3
  Grade 1-2 diverticulitis | 1
  Grade 3-4 sepsis | 1
  Grade 1-2 urinary tract infection | 1
  Grade 1-2 bruising | 1
  Grade 1-2 radiation recall reaction (dermatologic) | 1
  Grade 1-2 alanine aminotransferase increased | 4
  Grade 3-4 alanine aminotransferase increased | 2
  Grade 1-2 alkaline phosphatase increased | 4
  Grade 1-2 aspartate aminotransferase increased | 4
  Grade 3-4 aspartate aminotransferase increased | 1
  Grade 1-2 blood bilirubin increased | 1
  Grade 1-2 creatinine increased | 2
  Grade 1-2 hemoglobin increased | 1
  Grade 1-2 lymphocyte count decreased | 23
  Grade 3-4 lymphocyte count decreased | 13
  Grade 1-2 neutrophil count decreased | 22
  Grade 3-4 neutrophil count decreased | 24
  Grade 1-2 platelet count decreased | 21
  Grade 3-4 platelet count decreased | 1
  Grade 1-2 weight loss | 1
  Grade 3-4 weight loss | 1
  Grade 1-2 white blood cell decreased | 26
  Grade 3-4 white blood cell decreased | 26
  Grade 1-2 anorexia | 4
  Grade 3-4 hyperglycemia | 1
  Grade 1-2 hypermagnesemia | 1
  Grade 1-2 hypoalbuminemia | 1
  Grade 1-2 hypocalcemia | 1
  Grade 1-2 hypokalemia | 2
  Grade 1-2 hyponatremia | 1
  Grade 1-2 arthralgia | 6
  Grade 1-2 arthritis | 1
  Grade 1-2 back pain | 1
  Grade 1-2 bone pain | 1
  Grade 1-2 leg stiffness | 1
  Grade 1-2 muscle cramps | 1
  Grade 1-2 myalgia | 3
  Grade 1-2 neck pain | 1
  Grade 1-2 osteonecrosis of jaw | 1
  Grade 1-2 pain in extremity | 1
  Grade 1-2 dizziness | 4
  Grade 3-4 dizziness | 1
  Grade 1-2 dysgeusia | 5
  Grade 1-2 headache | 2
  Grade 1-2 spasticity | 1
  Grade 1-2 depression | 1
  Grade 1-2 insomnia | 3
  Grade 1-2 mood swings | 1
  Grade 1-2 breast pain | 1
  Grade 1-2 vaginal dryness | 1
  Grade 1-2 epistaxis | 2
  Grade 1-2 sore throat | 1
  Grade 1-2 voice alteration | 1
  Grade 1-2 alopecia | 19
  Grade 1-2 brittle nails | 1
  Grade 1-2 dry skin | 2
  Grade 1-2 hyperhidrosis | 3
  Grade 1-2 itchy skin | 3
  Grade 1-2 nail loss | 1
  Grade 1-2 oral fissure | 1
  Grade 1-2 rash acneiform | 1
  Grade 1-2 rash maculo-papular | 1
  Grade 1-2 hot flashes | 12
  Grade 1-2 hypertension | 2
  Grade 3-4 thromboembolic event | 1

7. Secondary Outcome: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: * PFS will be followed from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants-Kaplan Meier
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
percentage of participants-Kaplan Meier | 67.911 [52.934 to 79.025]

8. Secondary Outcome: Overall Response Rate (Complete Response + Partial Response)
Description: * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, dDisappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Time of progression (estimated to be 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
Participants | 18

9. Secondary Outcome: Clinical Benefit Rate (Complete Response + Partial Response + Stable Disease) for at Least 6 Months)
Description: * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, dDisappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Time of progression (estimated to be 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
Number analyzed (Participants) | 54
Participants | 45

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days following completion of treatment.
Arm/Group | Palbociclib + Letrozole or + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 3/54
Serious Adverse Events (participants affected / at risk) | 15/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole or + Fulvestrant (N=54)
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Death (General disorders) | 3
Fever (General disorders) | 1
Generalized weakness (General disorders) | 1
Cellulitis (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Superficial thrombophlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole or + Fulvestrant (N=54)
Anemia (Blood and lymphatic system disorders) | 43
Gout (Blood and lymphatic system disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 4
Blurred vision (Eye disorders) | 4
Cataract (Eye disorders) | 3
Dry eye (Eye disorders) | 2
Eye lid pain (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Red eye (Eye disorders) | 1
Watering eyes (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Broken tooth (Gastrointestinal disorders) | 2
C. difficile (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 30
Dry lips (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 20
Dysphagia (Gastrointestinal disorders) | 5
Gastric ulcer (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 29
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 17
Breast pain (General disorders) | 4
Buttock pain (General disorders) | 3
Chills (General disorders) | 13
Cold sensitivity (General disorders) | 1
Cold sweats (General disorders) | 1
Common cold (General disorders) | 4
Dilation of appendix with periappendiceal fat stranding seen on CT (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 18
Edema trunk (General disorders) | 2
Fatigue (General disorders) | 33
Fever (General disorders) | 9
Flu-like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 1
Generalized weakness (General disorders) | 1
Groin pain (General disorders) | 1
Intrascapular pain (General disorders) | 1
Leg pain (General disorders) | 1
Localized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 14
Wrist pain (General disorders) | 1
Allergic reaction (Immune system disorders) | 3
Bladder infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 5
Diverticulitis (Infections and infestations) | 1
Fungal toe infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory syncytial virus (RSV) (Infections and infestations) | 1
Rhinovirus (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 9
Skin infection (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 7
Vaginal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Yeast infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Bug bite (Injury, poisoning and procedural complications) | 3
Burn (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 11
Fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Puncture wound (Injury, poisoning and procedural complications) | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Snake bite (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 18
Alkaline phosphatase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 19
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 18
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 40
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 47
Platelet count decreased (Investigations) | 23
Weight gain (Investigations) | 1
Weight loss (Investigations) | 6
White blood cell count decreased (Investigations) | 52
Anorexia (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 17
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 17
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 6
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 17
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 19
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 16
Back spasms (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Knee pain (Musculoskeletal and connective tissue disorders) | 3
Leg stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Sacroliac joint pain (Musculoskeletal and connective tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 20
Dysgeusia (Nervous system disorders) | 11
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 21
Memory impairment (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 9
Right arm numbness (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 2
Spasticity (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 9
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 11
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 20
Mood swings (Psychiatric disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 2
Vaginal itching (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
COPD (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Nasal drainage (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 22
Bilateral nares sores (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Brittle nail (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Erythema right breast (Skin and subcutaneous tissue disorders) | 1
Fever blister (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7
Itchy skin (Skin and subcutaneous tissue disorders) | 3
Nail loss (Skin and subcutaneous tissue disorders) | 1
Oral fissure (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculopapular (Skin and subcutaneous tissue disorders) | 10
Shoulder nodule (Skin and subcutaneous tissue disorders) | 1
Skin bump (Skin and subcutaneous tissue disorders) | 2
Stomach rash (Skin and subcutaneous tissue disorders) | 1
Tender nail bed (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 21
Hypertension (Vascular disorders) | 36
Lymphedema (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03007979/Prot_SAP_000.pdf